CLINICAL TRIAL: NCT03281096
Title: A Randomized Trial of Berberine Hydrochloride to Prevent Colorectal Adenomas in Patients With Previous Colorectal Cancer
Brief Title: A Research of Berberine Hydrochloride to Prevent Colorectal Adenomas in Patients With Previous Colorectal Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, xiaohua li, Director of colorectal surgery center, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJLL 2016 001
Record Dates: First submitted 2017-08-30; First posted 2017-09-13 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Adenomas

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine hydrochloride group (Experimental): Berberine hydrochloride 300mg tablet by mouth, two times per day for 3 years
  Interventions: Drug: Berberine hydrochloride
- Placebo (Placebo Comparator): identical-appearing placebo 300mg tablet by mouth, two times per day for 3 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berberine hydrochloride — patients take the Berberine hydrochloride 300mg tablet by mouth, 2 times a day with 3 years.
  Other Names: Berberine hydrochloride tablet ("Sine Tianping")
  Arms: Berberine hydrochloride group
Drug: Placebo — pill manufactured to mmic Berberine hydrochloride 100mg tablet
  Other Names: Placebo (for Berberine hydrochloride)
  Arms: Placebo

SUMMARY:
Experimental studies in animals and observational studies in humans suggest that fusobacterium nucleatum is associates with stages of colorectal neoplasia development, and Berberine Hydrochloride could rescue Fusobacterium nucleatum-induced colorectal tumorigenesis by modulating the tumor microenvironment. Whether regular Berberine Hydrochloride use may decrease the risk of colorectal adenomas, the precursors to most colorectal cancers is worth to further study.

DETAILED DESCRIPTION:
The prevalence of colorectal adenomas is high in our country, as is the incidence of colorectal cancer. It is well-known that colorectal adenomas are the precursor of colorectal cancer and that removing them will prevent colorectal cancer. Because most colorectal cancers arise from benign adenomas, adenomas have been used as surrogate end points in prevention trials. Berberine hydrochloride, which is an alkaloid extracted from Rhizoma coptidis, has been traditionally used in Chinese medicine to treat gastrointestinal infections, due to its antimicrobial properties. Previous clinical research and animal studies have demonstrated the anti-tumor action of Berberine hydrochloride. Persons with a history of colorectal cancer might constitute a group at higher risk for adenomas and thus be particularly suitable for a study of the chemopreventive effects of Berberine hydrochloride. Here, a randomized, double-blind, placebo-controlled trial was designed to determine whether the daily use of 300 mg of berberine hydrochloride could decreases the occurrence of new colorectal adenomas among patients with a history of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* Patients who had histologically documented colon or rectal cancer with a low risk of recurrent disease
* Patients with Dukes' stage A or B1 colon or rectal cancer (tumor-node-metastasis [TNM] stage T1 to T2, N0, M0) who had undergone curative resection of the primary tumor were immediately eligible for enrollment
* Patients with Dukes' stage B2 or C (T3 to T4, N0 to N1, M0) colon or rectal cancer who had undergone curative resection of the primary tumor were eligible if they had been free of disease for more than five years after curative surgery
* Eligible participants had to have undergone, after adequate preparation, colonoscopy to the cecum (or small-bowel anastomosis), with removal of all polyps, within four months before study entry
* Patients were eligible if they were in good general health, with an expected survival of at least five years; willing to provide and able to understand informed consent and to cooperate with the study procedures; not currently enrolled in a clinical trial of colon-cancer treatment or other chemoprevention trial; and not pregnant or nursing.

Exclusion Criteria:

* Patients who are hypersensitive or intolerant to the drugs
* Patients had familial polyposis
* Patients had invasive cancer other than nonmelanoma skin cancer within 5 years before the intake appointment
* Patients with diabetes mellitus, severe renal disease or cardiovascular disease (defined by a New York Heart Association functional classof III or IV)
* Patients with hypercalcemia or urolithiasis
* Patients had a history of inflammatory bowel disease
* Patients with hemolytic anemia and glucose -6- phosphate dehydrogenase deficiency
* Patients had received immunosuppressive therapy within the previous 6 months
* Patients had clinically obvious narcotic or alcohol dependence during the previous 6 months
* Patients had used NSAIDs including aspirin at any dose on 3 or more days per month during each of the 3 months before enrollment or for a period of 36 days in the previous year; or had a history of stroke, transient ischemic attacks, angina, myocardial infarction, or atherosclerotic peripheral vascular disease
* Pregnant women, women during breast-feeding period, or women with expect pregnancy
* Patients with a history of subtotal gastrectomy or partial bowel resection
* Patients who are not able to cooperate
* Patients with any condition that could be worsened by supplemental Berberine hydrochloride

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Cumulative the colorectal adenoma incidence rate during Berberine hydrochloride or placebo treatment in patients with a history of colorectal cancer | From baseline to 3 years.
  The proportion of patients in whom one or more colorectal adenomas were investigated during the period from one year after randomization through the anticipated surveillance follow-up examination. The development of colorectal adenomas was assessed with an Olympus flexible video colonoscopy. One endoscopic investigator, who did not review the records of previous examinations, made all the assessments.

SECONDARY OUTCOMES:
Cumulative the numbers or diameters of those new colorectal adenomas during Berberine hydrochloride or placebo treatment in patients with a history of colorectal cancer | From baseline to 3 years.
  The numbers or diameters of those new colorectal adenomas were analyzed during the period from one year after randomization through the anticipated surveillance follow-up examination. The endoscopic investigator, who did not review the records of previous examinations, counted the total number of colorectal adenomas, and the examination was recorded on videotape. The diameter of those colorectal adenomas was measured in millimeters with a graduated scale passed through the colonoscopy biopsy channel.

CONTACTS AND LOCATIONS:
Overall Officials: Weizhong Wang, MD,PH.D, Principal Investigator — Xijing digestive surgery center
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China